CLINICAL TRIAL: NCT01995630
Title: Optical Quality After Implantation of a Spherical or Aspherical Intraocular Lens in Hypermetropic Patients: A Randomized Clinical Trial
Brief Title: Optical Quality After Implantation of a Spherical or Aspherical Intraocular Lens in Hypermetropic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Navid Ardjomand, Univ.-Doz. Dr. med. univ., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIOLvsAIOL
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Cataract; Spherical Aberrations; Intraocular Lenses; Depth of Focus
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hypermetropic, spherical IOL (Experimental): AMO Sensar AR40e
  Interventions: Device: AMO Sensar AR40e
- Hypermetropic, aspheric IOL (Experimental): AMO Tecnis ZA9003
  Interventions: Device: AMO Tecnis ZA9003
- Emmetropic, spherical IOL (Active Comparator): AMO Sensar AR40e
  Interventions: Device: AMO Sensar AR40e
- Emmetropic, aspheric IOL (Active Comparator): AMO Tecnis ZA9003
  Interventions: Device: AMO Tecnis ZA9003

INTERVENTIONS:
Device: AMO Tecnis ZA9003
  Arms: Emmetropic, aspheric IOL; Hypermetropic, aspheric IOL
Device: AMO Sensar AR40e
  Arms: Emmetropic, spherical IOL; Hypermetropic, spherical IOL

SUMMARY:
The purpose of this study is to evaluate differences in the depth of focus after implantation of a spherical or aspheric IOL in hypermetropic and emmetropic patients. After implantation of a spherical IOL hypermetropic patients may achieve a better depth of focus compared to emmetropic patients due to a larger amount of spherical aberrations.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Dioptric power of IOL >22.0 D in hypermetropic patients and 18.0-22.0 D in emmetropic patients, respectively

Exclusion Criteria:

* Uveitis, pathology of the retina or the optic nerve
* Corneal scarring or irregularities
* Astigmatism >1.5 D
* Amblyopia
* Perioperative complications
* Postoperative refractive error >2.0 D of spherical equivalent
* Postoperative DCVA <0.8 (ETDRS)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06-26 (Actual)

PRIMARY OUTCOMES:
Distance-corrected intermediate visual acuity | 3 month postop

SECONDARY OUTCOMES:
Distance-corrected near visual acuity | 3 month postop
Uncorrected distance visual acuity | 3 month postop
Corrected distance visual acuity | 3 month postop
Uncorrected near visual acuity | 3 month postop
Corrected near visual acuity | 3 month postop
Pseudoaccomodation | 3 month postop
Photopic contrast sensitivity | 3 month postop
Mesopic contrast sensitivity | 3 month postop
Spherical aberrations | 3 month postop
High order aberrations | 3 month postop

CONTACTS AND LOCATIONS:
Overall Officials: Navid Ardjomand, MD, Principal Investigator — Dept. of Ophthalmology, Medical University of Graz
Locations (1):
- Dept. of Ophthalmology, Medical University of Graz, Graz, Austria